CLINICAL TRIAL: NCT07152886
Title: The Effects of Clostridium Butyricum on Adverse Events During Adjuvant Chemotherapy for Colorectal Cancer: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Trial
Brief Title: The Effects of Clostridium Butyricum on Adverse Events During Adjuvant Chemotherapy for Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Linyi People's Hospital (Other); Shandong Cancer Hospital and Institute (Other); Yantai Yuhuangding Hospital (Other); Jining First People's Hospital (Other); Rizhao People's Hospital (Other); Qianfoshan Hospital (Other); Weifang People's Hospital (Other); Qilu Hospital of Shandong University (Other); Taian City Central Hospital (Other); The Affiliated Hospital of Shandong Second Medical University (Unknown); Dongying People's Hospital (Other)
Responsible Party: Principal Investigator, Zhou Yanbing, The Director of the Department of Gastrointestinal Surgery, the Affiliated Hospital of Qingdao University, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DHQDFY-02
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer; Chemotherapeutic Toxicity
Keywords: Colorectal Cancer; adjuvant chemotherapy; Clostridium butyricum
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Eligible participants who meet the inclusion criteria after screening will receive either the investigational product or placebo, packaged and labeled with a unique randomization number, as assigned by an independent investigator. The participants, as well as the researchers involved in recruitment, screening, and follow-up, and the nursing staff, will all be blinded to the group assignments. Unblinding and data analysis will be conducted only after all participants have completed adjuvant chemotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Oral administration of Clostridium butyricum capsules during adjuvant chemotherapy, 6 capsules tid. (each capsule containing ≥6.3 × 10⁶ CFU of Clostridium butyricum).
  Interventions: Drug: Clostridium butyricum capsules
- control group (Placebo Comparator): Oral administration of placebo capsules, 6 capsules three times daily, containing corn starch. The appearance and weight of the placebo capsules are identical to those of intervention group.
  Interventions: Other: placebo capsules

INTERVENTIONS:
Drug: Clostridium butyricum capsules — Clostridium butyricum capsules , 6 capsules tid (each capsule containing ≥6.3 × 10⁶ CFU of Clostridium butyricum).
  Arms: intervention group
Other: placebo capsules — Oral administration of placebo capsules, 6 capsules tid., containing corn starch. The appearance and weight of the placebo capsules are identical to those of intervention group.
  Arms: control group

SUMMARY:
This study is a multicenter randomized controlled trial designed to investigate the effects of Clostridium butyricum on adverse events during adjuvant treatment for colorectal cancer.

DETAILED DESCRIPTION:
A total of 238 participants who have undergone radical resection for colorectal cancer and are scheduled to initiate adjuvant chemotherapy will be enrolled and randomly assigned in a 1:1 ratio to the intervention group or the control group. During adjuvant chemotherapy, participants in the intervention group will receive Clostridium butyricum capsules, while those in the control group will receive a placebo. The primary outcome is the incidence of CTCAE grade 3-4 diarrhea during adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years;
* No restriction on gender;
* Have completed radical resection for colorectal cancer (including open, laparoscopic, or robotic surgery), and assessed by the MDT as requiring adjuvant therapy primarily based on 5-FU and its derivatives or platinum-based regimens (including chemotherapy, targeted therapy, or radiotherapy);
* ECOG performance status score of 0-2;
* Signed informed consent

Exclusion Criteria:

* Use of probiotics, prebiotics, synbiotics, or antibiotics within 2 weeks prior to enrollment;
* Presence of psychiatric disorders or other conditions that prevent cooperation with the intervention;
* Dysfunction of vital organs such as the liver, kidneys, or heart that renders the individual unsuitable for clinical research upon assessment, or inadequate bone marrow, liver, or renal function to undergo adjuvant therapy;
* Participation in other clinical studies within 3 months prior to enrollment;
* History of inflammatory bowel disease;
* History of autoimmune diseases;
* Pregnancy or breastfeeding;
* Receipt of neoadjuvant therapy (including chemotherapy, radiotherapy, or targeted therapy) prior to surgery;
* Underwent ostomy surgery during the operation (including temporary or permanent ostomy).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
CTCAE grade 3-4 diarrhea | Throughout the entire course of adjuvant chemotherapy , up to 6 months
  Incidence of grade 3-4 diarrhea during adjuvant chemotherapy, with severity graded according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0

SECONDARY OUTCOMES:
Overall incidence of adverse events | Throughout the entire course of adjuvant chemotherapy , up to 6 months
  Overall incidence of adverse events during adjuvant chemotherapy. Severity and specific types will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
rate of adjuvant treatment interruption | Throughout the entire course of adjuvant chemotherapy , up to 6 months
  defined as a delay of >=3 weeks from the planned treatment schedule
White blood cell count | Before the start of each cycle of adjuvant chemotherapy. A total of 6 to 8 cycles of chemotherapy are expected to be administered.
  Blood samples will be collected and tested before the start of each cycle of adjuvant chemotherapy to obtain the results.
neutrophil count | Before the start of each cycle of adjuvant chemotherapy. A total of 6 to 8 cycles of chemotherapy are expected to be administered.
  Blood samples will be collected and tested before the start of each cycle of adjuvant chemotherapy to obtain the results.
lymphocyte count | Before the start of each cycle of adjuvant chemotherapy. A total of 6 to 8 cycles of chemotherapy are expected to be administered.
  Blood samples will be collected and tested before the start of each cycle of adjuvant chemotherapy to obtain the results.
C-reactive protein | Before the start of each cycle of adjuvant chemotherapy. A total of 6 to 8 cycles of chemotherapy are expected to be administered.
  Blood samples will be collected and tested before the start of each cycle of adjuvant chemotherapy to obtain the results.
procalcitonin | Before the start of each cycle of adjuvant chemotherapy. A total of 6 to 8 cycles of chemotherapy are expected to be administered.
  Blood samples will be collected and tested before the start of each cycle of adjuvant chemotherapy to obtain the results.
serum albumin | Before the start of each cycle of adjuvant chemotherapy. A total of 6 to 8 cycles of chemotherapy are expected to be administered.
  Blood samples will be collected and tested before the start of each cycle of adjuvant chemotherapy to obtain the results.
serum procalcitonin | Before the start of each cycle of adjuvant chemotherapy. A total of 6 to 8 cycles of chemotherapy are expected to be administered.
  Blood samples will be collected and tested before the start of each cycle of adjuvant chemotherapy to obtain the results.
completion rate of the planned adjuvant therapy | Throughout the entire course of adjuvant chemotherapy , up to 6 months
  The total number of adjuvant chemotherapy cycles will be determined by the MDT (Multidisciplinary Team) prior to the initiation of treatment. Completion of the planned number of cycles as specified will be defined as "completed."

CONTACTS AND LOCATIONS:
Overall Officials: Yanbing Zhou, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No